CLINICAL TRIAL: NCT05202314
Title: Camrelizumab Combined With Neoadjuvant Chemotherapy After Stent Placement Versus Surgery Alone for Left-Sided Obstructive Colonic Cancer
Brief Title: Camrelizumab Combined With Neoadjuvant Chemotherapy After Stent Placement for Left-Sided Obstructive Colonic Cancer
Acronym: NACSOC-02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Professor, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12-24
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer; Neoadjuvant Chemotherapy; Stent; Obstruction; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Bites and Stings | interventions — Immunotherapy; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy group (Experimental): After clinical success of colonic stenting, regardless of the MSI state all patients will receive Immunotherapy (Camrelizumab 200mg) for 2 cycles compined with neoadjuvant chemotherapy with mFOLFOX6 regimen for 3 cycles or CapeOx regimen for 2 cycles. Patients will undergo surgery 2-3 weeks after the last cycle of chemotherapy, type and extent of the surgery will be selected by the surgeon.
  Interventions: Drug: Immunotherapy (Camrelizumab)

INTERVENTIONS:
Drug: Immunotherapy (Camrelizumab) — After clinical success of colonic stenting, regardless of the MSI state, patients will receive Immunotherapy (Camrelizumab 200mg) for 2 cycles compined with neoadjuvant chemotherapy with mFOLFOX6 regimen for 3 cycles or CapeOx regimen for 2 cycles. Patients will undergo surgery 2-3 weeks after the last cycle chemotherapy
  Other Names: Chemotheray (CAPOX or mFOLFOX6)

SUMMARY:
Patients with obstruction are associated with worse oncologic outcomes compared with those having nonobstructive tumors. Conventionally, patients with malignant large bowel obstruction receive emergency surgery, with morbidity rates of 30%-60% and mortality rates of 7-22%, and about two-thirds of such patients end up with a permanent stoma. Self-expanding metallic stents (SEMS) haven been used as a bridge to surgery (to relieve obstruction prior to elective surgery) in patients with potentially resectable colorectal cancer. Several clinical trials demonstrate that SEMS as a bridge to surgery may be superior to emergency surgery considering the short-term outcomes. SEMS is associated with lower morbidity and mortality rate, increased primary anastomosis rate, and decreased stoma creation rate. Although about half of patients can achieve primary anastomosis after stent placement, the primary anastomosis rate is still significantly lower compared with nonobstructing elective surgery. The interval between stent placement and surgery may be not long enough that bowel decompression is insufficient at the time of operation. Furthermore#the long-term oncologic results regarding SEMS as a bridge to surgery are still limited and contradictory. Sabbagh et al. suggest worse overall survival of patients with SEMS insertion compared with emergency surgery, the 5-year cancer-specific mortality was significantly higher in the SEMS group (48% vs 21%, respectively, P=0.02). One interpretation is that tumor cells may disseminate during the procedure of colonic stenting placement. Immunotherapy has proven to be highly effective as first-line treatment of metastatic colorectal cancer (CRC). And immunotherapy also has emerged as a neoadjuvant approach, possibly changing treatment strategy for both primary resectable and metastatic CRC. We hypothesis that, regardless of the MSI state, immunotherapy (Camrelizumab, an anti-PD-1 antibody) combined with chemotherapy after stenting may improve overall survival by eradicating micrometastasis. Moreover, immunotherapy (Camrelizumab, an anti-PD-1 antibody) combined with neoadjuvant chemotherapy prolongs the interval between stent placement and surgery, and the time for bowel decompression is more sufficient, which may increase the success rate of primary anastomosis and decrease risk of stoma formation, and furthermore, improve OS and PFS.

DETAILED DESCRIPTION:
We hypothesis that, regardless of the MSI state, immunotherapy combined with immediate chemotherapy after stenting may improve overall survival by eradicating micrometastasis. Moreover, immunotherapy (Camrelizumab, an anti-PD-1 antibody) combined with neoadjuvant chemotherapy prolongs the interval between stent placement and surgery, and the time for bowel decompression is more sufficient, which may increase the success rate of primary anastomosis and decrease risk of stoma formation, and furthermore, improve OS and PFS.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically proven colonic obstruction of the left colon/upper rectum presumed secondary to a carcinoma
* Able to give written, informed consent
* Primary tumor was resectable
* ECOG score 0 or 1
* Haemoglobin greater than 100 g/L after transfusion before chemotherapy,
* White blood cells greater than 3.0×10# /L
* Platelets greater than 100×10# / L;
* Glomerular filtration rate greater than 50 mL per minute as calculated by the Wright or Cockroft formula
* Bilirubin less than 1.5×Upper Limit of Normal(ULN)
* ALT and AST less than 2.5×ULN

Exclusion Criteria:

* Distal rectal cancers(equal or less than 10cm from the anal verge)
* Patients with signs of peritonitis and/or bowel perforation
* Patients who did not give informed consent
* Patients who were considered unfit for operative treatment or refuse surgery.
* Patients with suspected or proven metastatic adenocarcinoma;
* Patients with unresectable colorectal cancer, or planning for palliative treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission | 2 weeks after patients received radical operation
  No tumor cell found in surgical specimens

SECONDARY OUTCOMES:
Disease Free Survival | 3 years after operation
  No tumor regrowth or recurrence or metastasis found
Overall Survival | 3 years after operation
  Survive during following

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Jun Wang, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No